CLINICAL TRIAL: NCT01202825
Title: Phase I, First-in-human Trial in Healthy Volunteers to Examine Increasing Single and Repeated Oral Doses of TMC647055, Followed by a Repeated-dose Part in Chronic HCV-genotype 1 Infected Patients to Examine TMC647055 Given Alone or in Combination With TMC435
Brief Title: TMC647055HPC1001 - First-in-human Trial to Examine Safety, Tolerability and Pharmacokinetics (How the Drug is Absorbed Into the Bloodstream) of Increasing Single Oral Doses and of Increasing Repeated Oral Doses of TMC647055 in Healthy Volunteers and in Hepatitis C Virus Infected Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tibotec Pharmaceuticals, Ireland (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: CR017035; TMC647055HPC1001 (Other: Tibotec Pharmaceuticals, Ireland)
Record Dates: First submitted 2010-09-14; First posted 2010-09-16 (Estimated); Last update posted 2013-03-04 (Estimated); Status verified 2013-03

CONDITIONS: Hepatitis C
Keywords: HCV genotype 1 infected patients; TMC647055HPC1001; TMC647055; HPC; Hepatitis C; Healthy volunteers; TMC435
MeSH Terms: conditions — Hepatitis C | interventions — 27-cyclohexyl-12,13,16,17-tetrahydro-22-methoxy-11,17-dimethyl-10,10-dioxide-2,19-methano-3,7:4,1-dimetheno-1H,11H-14,10,2,9,11,17-benzoxathiatetraazacyclo docosine-8,18(9H,15H)-dione; Simeprevir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (10):
- 001 (Experimental)
  Interventions: Drug: TMC647055
- 008 (Placebo Comparator)
  Interventions: Drug: Placebo
- 002 (Placebo Comparator)
  Interventions: Drug: Placebo
- 009 (Experimental)
  Interventions: Drug: TMC647055
- 003 (Experimental)
  Interventions: Drug: TMC647055
- 004 (Placebo Comparator)
  Interventions: Drug: Placebo
- 005 (Experimental)
  Interventions: Drug: TMC647055
- 010 (Experimental)
  Interventions: Drug: TMC435
- 006 (Placebo Comparator)
  Interventions: Drug: Placebo
- 007 (Experimental)
  Interventions: Drug: TMC647055

INTERVENTIONS:
Drug: TMC647055 — One single dose as oral solution, doses from 100 mg up to a maximum of 3000 mg increasing in sessions I through VI.
  Arms: 001
Drug: Placebo — Oral solution given in session XI every 12 hours, in session XII every 12 or 8 hours. Doses and regimen will be determined based on outcome of previous sessions.
  Arms: 008
Drug: TMC647055 — Oral solution given in session XIII, treatment arm 1 during 10 days at a dose of 1000 mg every 12 hours.
  Arms: 009
Drug: TMC647055 — In sessions VIII through X, oral solution given once daily, every 12 hours or every 8 hours on 6 consecutive days. Doses are based on outcome of previous sessions.
  Arms: 005
Drug: Placebo — One single dose as oral solution, selected dose ranging between 100 and 3000 mg in session VII
  Arms: 002
Drug: TMC435 — Oral capsule given in session XIII, in treatment arm 1 during 10 days and in treatment arm 2 during 6 days at a dose of 150 mg once daily.
  Arms: 010
Drug: Placebo — One single dose as oral solution, selected dose ranging between 100 and 3000 mg in session VII
  Arms: 004
Drug: TMC647055 — One single dose as oral solution, selected dose ranging between 100 and 3000 mg in session VII
  Arms: 003
Drug: Placebo — In sessions VIII through X, oral solution given once daily, every 12 hours or every 8 hours on 6 consecutive days. Doses are based on outcome of previous sessions.
  Arms: 006
Drug: TMC647055 — Oral solution given in session XI every 12 hours, in session XII every 12 or 8 hours. Doses and regimen will be determined based on outcome of previous sessions.
  Arms: 007

SUMMARY:
The purpose of this study is to assess the safety and tolerability of TMC647055 both after increasing single oral doses from 100 mg up to maximum 3000 mg in fed conditions, and after multiple oral doses in fed conditions at increasing dose levels administered for 6 days, as well as to assess the pharmacokinetics of TMC647055 after increasing single oral doses from 100 mg up to maximum 3000 mg in fed conditions, and after multiple oral doses in fed conditions at increasing dose levels administered for 6 days and to assess the effect of food on a single oral dose of TMC647055 at one dose level, all in healthy participants. In addition, the safety, tolerability, pharmacokinetics and the antiviral activity of TMC647055 will be determined after 6 days of consecutive dosing and of TMC647055 and TMC435 after 10 days of co-administration in chronic hepatitis C virus infected patients. Pharmacokinetics means how the drug is absorbed into the bloodstream, distributed in the body and eliminated from the body. TMC647055 is being investigated for the treatment of chronic hepatitis C infection.

DETAILED DESCRIPTION:
TMC647055 is being investigated for the treatment of chronic hepatitis C infection. This is a first-in-human, double-blind (sponsor, investigator and participant do not know which treatment is given), randomized (like flipping a coin), placebo-controlled, single centre, Phase I study in healthy volunteers to examine the safety, tolerability, and plasma pharmacokinetics of increasing single oral doses and of increasing repeated oral doses of TMC647055, followed by a double-blind repeated-dose part in chronic hepatitis C virus (HCV) infected patients. The study population will consist of 45 healthy adult volunteers between 18 and 55 years of age and 10 or 20 chronic HCV-genotype 1 infected patients between 18 and 65 years of age. The single dose escalation part of the trial will include 2 panels (Panels 1 and 2) of 9 participants each. There will be 6 sessions (Sessions I to VI): panel 1 will do sessions I, III & V; panel 2 will do sessions II, IV and VI. In each session, 6 participants will receive TMC647055 and 3 participants will receive placebo with standard meals. Over 3 sessions, each participant will receive TMC647055 twice and placebo once. The dose of TMC647055 will be consecutively increased. Planned doses will be 100 mg, 250 mg, 600 mg, 1250 mg, 2000 mg, and 3000 mg of TMC647055 or placebo, administered as a single oral administration. A wash out period of at least 10 days will be respected between 2 sessions of 1 panel. Doses may be adapted pending the safety and pharmacokinetic outcome of the previous sessions but will not exceed the limit of 3000 mg. Dose increase will only occur if the previous dose is shown to be generally safe and tolerable. For precautionary safety reasons, the dose administration in sessions IV, V and VI will be staggered: the first 4 to 5 participants of the panel will receive the dose at least 24 hours prior to the second group of 4 to 5 participants. To investigate the effect of food, one single dose will be tested in fasted conditions (Session VII). The dose of TMC647055 tested in this session will be derived from the results obtained in Sessions I to V. Participants who received TMC647055 at the selected dose with standard meals in Sessions I to V will again receive TMC647055 in fasted conditions in Session VII. Participants who received placebo will receive placebo again. The multiple-dose escalation part of the trial (sessions VIII, IX and X) will include 3 panels (Panels 3, 4, and 5) of 9 participants each: panel 3 will do session VIII, panel 4 session IX and panel 5 session X. In all panels, TMC647055 or placebo will be administered during 6 consecutive days, with on Day 6 a morning dose only. Medication is anticipated to be given either every 8 hours, every 12 hours or every 24 hours. This can be changed per dosing session following the outcome of the previous session. In each multiple dosing session, 6 participants will receive TMC647055 and 3 participants will receive placebo. The multiple dose escalation part will be started when the doses of Sessions I, II, III, and IV are found to be generally safe and tolerable based upon review of the blinded safety and pharmacokinetic data. Dose increase will only occur if the previous dose is shown to be generally safe and tolerable. The initial daily dose tested in Panel 3 will not be higher than the doses tested in Sessions I to IV. After the healthy volunteer sessions, there will be 3 sessions in chronic HCV infected patients (sessions XI, XII and XIII). Session XI will be started when the doses in healthy volunteers are found to be generally safe and tolerable and a selected dose will be given every 12 hours. The total daily dose will not exceed the highest daily dose and exposure shown to be generally safe in the multiple dose escalation in healthy volunteers. The dose for session XII will be selected based on the results from session XI and will be given every 12 hours or every 8 hours. In each session, 8 patients will receive TMC647055 and 2 patients will receive placebo. TMC647055 will be given during 6 consecutive days with on day 6 a morning dose only. Session XIII will be open-label and will consist of 2 treatment arms. In treatment arm 1, 8 patients will receive TMC647055 (1000 mg twice a day) co-administered with TMC435 (150 mg once daily) for 10 days.In treatment arm 2, 8 subjects will receive TMC435 (150 mg once daily) for 6 days. Safety and tolerability will be evaluated continuously by checking illnesses and side effects, by taking blood and urine samples, by electrocardiograms and telemetry (electrical recording of the heart, only for healthy volunteers), by taking blood pressure and heart rate and by performing physical examinations. TMC647055 or placebo will be given as an oral solution, ranging from 100 to 3000 mg in the single dose part, in the multiple dose part during 6 consecutive days either every 8 hours, 12 hours or 24 hour. In sessions XI and XII, TMC647055 or placebo will be given every 8 or 12 hours at dose and frequency determined by results of the previous sessions. In session XIII, the dose of TMC647055 will be 1000 mg twice a day and TMC435 will be given as oral capsules at 150 mg once daily.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers should be healthy on the basis of physical examination, medical history, laboratory tests, triplicate electrocardiogram and vital signs, performed at screening, have a Body Mass Index (BMI, weight in kg divided by the square of height in meters) of 18.0 to 30.0 kg/m2, extremes included and be non-smoking for at least 3 months prior to selection
* Chronic hepatitis-C infected patients should have documented chronic genotype 1a or 1b HCV infection, otherwise no clinically relevant currently active disease and a BMI of 18.0 to 35.0 kg/m2, extremes included
* Women must be postmenopausal for at least 2 years, and/or be surgically sterile.

Exclusion Criteria:

* All participants with a drug allergy such as, but not limited to, sulfonamides and penicillins, or with a drug allergy as witnessed in previous trials with experimental drugs
* Use of concomitant medication, including over-the-counter products, herbal medication and dietary supplements, except for paracetamol (acetaminophen) or ibuprofen or hormone replacement therapy or for chronic hepatitis-C infected patients products that are not CYP3A4 inhibitors or inducers and stable use of methadone, in a period of 14 days before the first trial medication administration
* Any condition that, in the opinion of the investigator, would compromise the study or the well-being of the subject or prevent the subject from meeting or performing study requirements
* History or suspicion of current use of alcohol, barbiturate, amphetamine, recreational or narcotic drug use, which in the investigator's opinion would compromise subject's safety and/or compliance with the trial procedures
* Participation in an investigational drug trial or having received an investigational vaccine within 30 days prior to the first intake of TMC647055 or placebo.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2010-04; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
The number of participants with adverse events per type as a measure of safety and tolerability after increasing single and multiple oral doses in healthy volunteers. | Continuously from screening until the last follow-up visit 30 to 35 days after last drug intake.
Plasma and urine concentration of TMC647055 after increasing single and multiple oral doses in healthy volunteers in fed conditions. | For single dose sessions in plasma on days 1 (multiple times), 2 (2 times), 3 and 4 and continuous urine collection on days 1 and 2 of session IV only. For multiple dose sessions on days 1 and 6 multiple times, on day 7 2 times and on days 2-3-4-5-8-9.
Plasma concentration of TMC647055 after a single oral dose in healthy volunteers in fasted conditions as compaired to fed conditions. | For session 7, in plasma on days 1 (multiple timepoints), 2 (2 timepoints), 3 and 4.
Plasma concentration of TMC647055 after 6 days oral dosing in chronic HCV-genotype 1 infected patients. | On days 1 and 6 multiple times and on days 2-3-4-5-7-8-9 pre-dose.
The number of participants with adverse events per type as a measure of safety and tolerability after 6 days oral dosing in chronic HCV-genotype 1 infected patients. | Continuously from screening until the last follow-up visit 30 to 35 days after last drug intake.
Plasma concentration of TMC647055 after a single oral dose in healthy volunteers in fasted conditions as compared to fed conditions. | For session 7, in plasma on days 1 (multiple timepoints), 2 (2 timepoints), 3 and 4.
The number of participants with adverse events per type as a measure of safety and tolerability after 6 days of TMC647055, after 10 days co-administration of TMC647055 and TMC435 and after 6 days of TMC435 in chronic HCV-genotype 1 infected patients. | Continuously from screening until the last follow-up visit 30 to 35 days after last drug intake.
Plasma concentration of TMC647055 and TMC435, if applicable, in chronic HCV-genotype 1 infected patients. | Sessions XI and XII: on days 1 and 6 multiple times and on days 2-3-4-5-7-8-9 pre-dose. Session XIII: on days 1, 6 and 10 (if applicable) multiple times and on other days pre-dose.

SECONDARY OUTCOMES:
HCV RNA decrease will be measured at the tested dose(s) and regimen(s) in chronic HCV-genotype 1 infected patients. | At screening, day 1 through day 9 at several timepoints.
HCV RNA will be measured in chronic HCV-genotype 1 infected patients. | Session XI and XII: at screening, day 1 through day 9 at several timepoints. Session XIII: at screening, day 1 through day 10 (TMC435 alone) or 14 (co-administration) at several timepoints and at the 3 follow-up visits.

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec Pharmaceuticals Clinical Trial, Study Director — Tibotec Pharmaceutical Limited
Locations (1):
- Antwerp, Belgium